CLINICAL TRIAL: NCT06571149
Title: Safety and Efficacy of Intravenous Thrombolysis in Patients With Ischemic Stroke on Treatment With Direct Oral Anticoagulants: DO-IT - The DOAC Intravenous Thrombolysis Trial
Brief Title: Safety and Efficacy of Intravenous Thrombolysis in Patients With Ischemic Stroke and Direct Oral Anticoagulants Intake
Acronym: DO-IT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01157
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: DOAC; NOAC (Novel Oral Anticoagulants); Anticoagulation; r-tPA (tissue-type plasminogen activator); Alteplase; Tenecteplase; Rivaroxaban; Apixaban; Dabigatran; Edoxaban
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Medical Treatment (standard of care) (No Intervention): Patients will receive Standard of care/Best medical treatment according to local applicable guidelines, including the current American Heart Association/American Stroke Association (AHA/ASA) and European Stroke Organisation/ European Society of Minimally Invasive Neurological Therapy (ESO/ESMINT) guidelines.
- Intravenous Thrombolysis + Best medical treatment (standard of care) (Experimental): Patients will receive intravenous administration of Tenecteplase or Alteplase.
  Interventions: Drug: Tenecteplase or Alteplase

INTERVENTIONS:
Drug: Tenecteplase or Alteplase — Patients randomized to intravenous thrombolysis (IVT) treatment will receive intravenous Tenecteplase or Alteplase.
  Arms: Intravenous Thrombolysis + Best medical treatment (standard of care)

SUMMARY:
DO-IT is an international, multicenter, prospective, two-arm, randomized, open label, blinded endpoint superiority trial determining the safety and efficacy of intravenous thrombolysis (IVT) in participants experiencing an acute ischemic stroke (AIS) with recent (within the last 48 hours) intake of direct oral anticoagulant (DOAC). For this purpose, 906 adult participants experiencing an AIS with recent DOAC intake will be enrolled at several high-volume international stroke centers and randomly assigned in a ratio of 1:1 to one of two treatment arms: (1) IVT and standard of care/best medical treatment or (2) standard of care/best medical treatment. The DO-IT trial is a definitive test of the hypothesis that IVT is superior to standard of care for achieving better outcome at 90 days in AIS participants with recent DOAC intake.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent (deferred consent when possible according to national legislation)
* AIS eligible to receive intravenous alteplase/tenecteplase as per standard of care disabling according to the judgement of the treating physician
* DOAC ingestion within 48 hours prior to enrollment, or patient with an ongoing prescription of DOAC but exact time point of last intake is unknown.
* Either

  * Can be randomized within 4 hours 15 minutes and treated within 4 hours 30 minutes of last known well time OR
  * MRI showing a pattern of "DWI-FLAIR-mismatch", i.e. acute ischemic lesion visibly on DWI ("positive DWI") but no marked parenchymal hyperintensity visible on FLAIR ("negative FLAIR") indicative of an acute ischemic lesion ≤4.5 hours of age AND Treatment can be started within 4.5 hours of symptom recognition (e.g., awakening).

Exclusion Criteria:

* Contra-indications to IVT by the current standard of care of the treating physicians with the exception of recent DOAC intake as specified above.
* Intended reversal by specific or unspecific reversal agents
* Pregnancy or lactating women. To be reasonable sure to exclude women with ongoing pregnancy, women are not considered of childbearing potential if they fulfill the following criteria

  * Age > 55 years OR
  * Age < 55 years and at least 12 months since last menstrual period OR
  * Have had a documented surgical sterilization
* Patient < 18 years of age (since the benefit of IVT is unproven in this population)

Since the benefit of IVT might be smaller in patients in which additional endovascular treatment is planned, the investigators will cap patients with intended mechanical thrombectomy at 20% of the trial population. If this number is reached, the following additional exclusion criterion will be applied:

* Intended treatment with endovascular reperfusion strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days +/- 2 weeks after randomization
  Modified Rankin Scale is a scale that runs from 0-6, running from perfect health without symptoms (0) to death (6).

SECONDARY OUTCOMES:
Dichotomized modified Rankin Scale (mRS) 0-2 (good functional outcome) | 90 days +/- 2 weeks post-randomization
  Modified Rankin Scale is a scale that runs from 0-6, running from perfect health without symptoms (0) to death (6).
Change from baseline in stroke severity (National Institutes of Health Stroke Scale, NIHSS) | 24 +/- 12 hours after Intervention
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. Thus, 0 (minimum score) means "no symptoms", whereas 42 (maximum score) means "severe stroke".
Health-related Quality of Life (EuroQol 5D-3L questionnaire) | 90 days +/- 2 weeks post-randomization
  The EuroQol 5D-3L (EuroQol 5 Dimensions with each 3 Levels) measures health-related Quality of Life.

OTHER OUTCOMES:
Rate of Symptomatic intracranial hemorrhage | Within the first 36 hours post-randomization
  Observed in clinical imaging
Rate of Major extracranial bleeding | Within the first 24 hours post-randomization
  Defined as clinically overt bleeding that is accompanied by one or more of the following (according to International Society on Thrombosis and Haemostasis definitions):
  * Decrease in haemoglobin of ≥ 2g / dl over a 24-hour period
  * Transfusion of ≥ 2 units of packed red blood cells
  * Occurring in a critical part of the body (intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, retroperitoneal)
  * In order for bleeding (e.g. gastrointestinal) in a critical area or organ to be classified as a major extracranial bleeding it must be associated with a symptomatic clinical presentation.
All-cause mortality | Up to 7 to 10 days after admission or until discharge, usually 2 weeks after admission
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meinel, MD, PhD, Study Director — Insel Gruppe AG, University Hospital Bern
Locations (14):
- UZ Leuven, Leuven, Belgium
- Hamilton Health Sciences, Hamilton, Ontario, Canada
- GHU Paris Psychiatrie et Neurosciences, Sainte Anne, Paris, France
- Heidelberg University Hospital, Heidelberg, Germany
- "Attikon" University Hospital, Athens, Greece
- National Cerebral and Cardiovascular Center Osaka, Osaka, Kansai, Japan
- Academic Medical Center Amsterdam, Department of Neurology, Amsterdam, Netherlands
- Canterbury District Health Board, Christchurch, New Zealand
- Akershus Hospital, Oslo, Norway
- Lisbon Central University Hospital Centre, Lisbon, Portugal
- Vall d'Hebron Stroke Center, Barcelona, Spain
- Switzerland (3):
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
IPDMA (individual participant data meta-analysis) of similar interventional clinical studies is planned.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of primary study results
Access Criteria: Ethics clearance, agreement with the DO-IT collaboration about terms of use and authorship